CLINICAL TRIAL: NCT06569212
Title: Beta-1 Adrenergic Inhibition to Reduce Cardiac Injury and Inflammation After Subarachnoid Hemorrhage (BADCATS)
Acronym: BADCATS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Madeleine Puissant (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Madeleine Puissant, Assistant Professor of Emergency Medicine, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2146714
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Non-Traumatic Subarachnoid Hemorrhage
Keywords: Beta-adrenergic blockade; Cardiac dysfunction; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoprolol (Beta-adrenergic blockade) (Experimental): Patients will receive metoprolol during the first 72-hours of hospitalization after non-traumatic SAH.
  Interventions: Drug: Metoprolol
- Placebo (Placebo Comparator): Patients will receive placebo during the first 72-hours of hospitalization after non-traumatic SAH.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol — Metoprolol Dosing:
  Metoprolol Injection (instructions: 5mg, once) Metoprolol Tab (25mg PO, q12 hours, timed to start 1hr after Metoprolol Injection, 6 doses) If unable to take PO medication, Metoprolol Injection (instructions, 5mg q6hrs for 12 doses) Continue for 72-hours of administration unless reaching stopping criteria
  Other Names: Metoprolol succinate
  Arms: Metoprolol (Beta-adrenergic blockade)
Drug: Placebo — Placebo Dosing:
  Placebo Injection (instructions: 5mL NS, once) Placebo Tab (1 tab PO, q12 hours, timed to start 1hr after placebo injection, 6 doses) If unable to take PO medication, Placebo Injection (instructions, 5mL q6hrs for 12 doses) Continue for 72-hours of administration unless reaching stopping criteria
  Arms: Placebo

SUMMARY:
To determine the effect of early metoprolol administration after non-traumatic subarachnoid hemorrhage (SAH).

DETAILED DESCRIPTION:
To determine the effect of early metoprolol administration after non-traumatic subarachnoid hemorrhage (SAH) on the brain and cardiac tissue damage and inflammation, we will conduct a pilot randomized controlled trial comparing (1) sympathetic nervous system (SNS) activation, (2) cardiac rhythm abnormalities, (3) biomarkers of brain and cardiac tissue damage, and (4) and neutrophil activity in patients receiving metoprolol (n=10) or placebo (n=10) for the first 72-hours after SAH.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Neuro-imaging confirmed non-traumatic subarachnoid hemorrhage

Exclusion Criteria:

* Traumatic cause of subarachnoid hemorrhage (e.g. fall, motor vehicle accident, other blunt trauma) as this is a different mechanism of hemorrhage.
* Other forms of traumatic or non-traumatic intracranial bleed including intracerebral hemorrhage (ICH), subdural hemorrhage, epidural hemorrhage
* Pregnancy (as the study medication, metoprolol, has FDA Pregnancy Category C rating)
* Unstable vital signs not amenable to beta-1 adrenergic receptor inhibitor (B1ARi) administration including:
* Systolic blood pressure < 80 mmHg not stabilized on vasopressor medications
* Heart rate < 50 bpm associated with hypotension
* Patients requiring vasopressor agents due to hypotension (SBP <80 mmHg)
* Other vital sign exclusion at the discretion of the treatment team
* Previous history of severe heart failure (Stage C or D Heart Failure and/or NYHA Class III or IV)
* Patient or legally authorized representative unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Delta QTc length | 7 days
  Change (Delta) QTc length between intervention and control groups.
Delta neutrophil activity | 7 days
  Delta neutrophil activity between intervention and control groups.

SECONDARY OUTCOMES:
Adverse events | 7-days
  Including but not limited to symptomatic bradycardia, symptomatic hypotension, or complete heart block
Number of patients with evidence of cardiac injury | 7-days
  Measurement of troponin levels, echocardiograph
Need for Vasopressors | 7-days
  Any documented intravenous vasoactive medication administration
Sympathetic Nervous System (SNS) Activity | 7-days
  Catecholamine Measurements
Neutrophil Activity | 7 days
  Measurement of neutrophils in CSF and serum samples
Evidence of Clinical Vasospasm | Up to 15-weeks
  Evidence of clinical vasospasm
ICU Length of Stay (LOS) | Up to 15-weeks
  Number of full days
Hospital Length of Stay (LOS) | Up to 15-weeks
  Number of full days
In-hospital mortality | Up to 15-weeks
  Whether patient died during during sentinel hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Puissant, MD, PhD, Principal Investigator — MaineHealth
Locations (1):
- MaineHealth, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study completion and until 6-months post-publication.
Access Criteria: A de-identified data set will be made available and people may request access to this.